CLINICAL TRIAL: NCT02284035
Title: Pilot 24week Clinical Trial to Assess the Safety, Tolerability and Efficacy of Dual Therapy With Raltegravir/Lamivudine Combination, Replacing Standard Combination Therapy in HIV-infected Pts With Prolonged Virological Suppression.
Brief Title: Safety & Efficacy of Dual Therapy With Raltegravir/Lamivudine
Acronym: RALAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Juan A. Arnaiz (Other)
Responsible Party: Sponsor-Investigator, Juan A. Arnaiz, Head Clinical Trials Unit, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RALAM; 2014-003142-27 (EudraCT Number)
Record Dates: First submitted 2014-10-28; First posted 2014-11-05 (Estimated); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 Raltegravir / 3TC (MK0518B (Experimental): Raltegravir / 3TC (MK0518B ) (50 patients)
  Interventions: Drug: Raltegravir/3TC
- Group 2 standard combination therapy (Active Comparator): NNRTI-Based Regimen:
  • EFV/TDF/FTC
  PI-Based Regimens:
  ATV/r + TDF/FTC or DRV/r + TDF/FTC
  INSTI-Based Regimens:
  DTG+ABC/3TC DTG+TDF/FTC EVG/cobi/TDF/FTC RAL+TDF/FTC
  NNRTI-Based Regimens:
  EFV plus ABC/3TC or RPV/TDF/FTC
  PI-Based Regimen:
  ATV/r plus ABC/3TC
  PI-Based Regimens:
  DRV/r + ABC/3TC or LPV/r + ABC/3TC or LPV/r + TDF/FTC
  INSTI-Based Regimen:
  RAL plus ABC/3TC
  And other ART regimens
  Interventions: Drug: EFV/TDF/FTC; Drug: ATV/r + TDF/FTC or DRV/r + TDF/FTC; Drug: DTG+ABC/3TC DTG+TDF/FTC EVG/cobi/TDF/FTC RAL+TDF/FTC; Drug: EFV plus ABC/3TC or RPV/TDF/FTC; Drug: ATV/r plus ABC/3TC; Drug: DRV/r + ABC/3TC or LPV/r + ABC/3TC or LPV/r + TDF/FTC; Drug: RAL plus ABC/3TC; Drug: Other ART regimens

INTERVENTIONS:
Drug: Raltegravir/3TC — MK0518B (Raltegravir/3TC) (300mg/150mg) twice daily, administered orally in the 300/150 mg film-coated tablets according to instructions in the prescribing information.
  Arms: Group 1 Raltegravir / 3TC (MK0518B
Drug: EFV/TDF/FTC — standard combination therapy
  Other Names: NNRTI-Based Regimen
  Arms: Group 2 standard combination therapy
Drug: ATV/r + TDF/FTC or DRV/r + TDF/FTC
  Other Names: PI-Based Regimens
  Arms: Group 2 standard combination therapy
Drug: DTG+ABC/3TC DTG+TDF/FTC EVG/cobi/TDF/FTC RAL+TDF/FTC
  Other Names: INSTI-Based Regimens
  Arms: Group 2 standard combination therapy
Drug: EFV plus ABC/3TC or RPV/TDF/FTC
  Other Names: NNRTI-Based Regimens
  Arms: Group 2 standard combination therapy
Drug: ATV/r plus ABC/3TC
  Other Names: PI-Based Regimen
  Arms: Group 2 standard combination therapy
Drug: DRV/r + ABC/3TC or LPV/r + ABC/3TC or LPV/r + TDF/FTC
  Other Names: PI-Based Regimens
  Arms: Group 2 standard combination therapy
Drug: RAL plus ABC/3TC
  Other Names: INSTI-Based Regimen
  Arms: Group 2 standard combination therapy
Drug: Other ART regimens
  Arms: Group 2 standard combination therapy

SUMMARY:
A pilot 24-week open-label, randomized, controlled clinical trial to assess the safety, tolerability and efficacy of dual therapy with Raltegravir/Lamivudine combination when replacing standard combination therapy in HIV-infected patients with prolonged virological suppression

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients will be males or females at least 18 years of age. Women of childbearing potential must have a negative pregnancy test within 10 days prior to randomization into the study.
2. Patients seropositive for HIV-1 using standard diagnostic criteria.
3. Patients virologically suppressed during at least 12 months prior to inclusion (viral load <50 copies/mL).
4. Patients on combination antiretroviral therapy (at least 2 antiretroviral drugs) for at least 12 months before being randomized in this study.
5. Patients who are clinically stable in the opinion of the investigator at study entry (clinical status and chronic medication must not have not been modified at least 14 days prior to randomization).
6. Patients who have signed informed consent to participate in the study.

Exclusion Criteria:

1. Pregnancy, lactation, or planned pregnancy during the study period.
2. Previous failure to an integrase inhibitor-containing regimen.
3. Previous failure to a 3TC or FTC-containing regimen.
4. Resistance mutations to 3TC or integrase inhibitor if any resistance test had been previously performed.
5. Any disease or history of disease which, in the opinion of the investigator, might confound the results of the study or pose additional risk to patient treatment.
6. Chronic hepatitis B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09-27 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Martinez, MD PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 75 participants were enrolled and randomized. One participant assigned to the Raltegravir/Lamivudine arm withdrew consent before starting treatment and was excluded from the analysis. As a result, 74 participants initiated treatment.
Groups:
- Group 1 Raltegravir / 3TC (MK0518B): Raltegravir / 3TC (MK0518B )
  Raltegravir/3TC: MK0518B (Raltegravir/3TC) (300mg/150mg) twice daily, administered orally in the 300/150 mg film-coated tablets according to instructions in the prescribing information.
- Group 2 Standard Combination Therapy: NNRTI-Based Regimen:
  • EFV/TDF/FTC
  PI-Based Regimens:
  ATV/r + TDF/FTC or DRV/r + TDF/FTC
  INSTI-Based Regimens:
  DTG+ABC/3TC DTG+TDF/FTC EVG/cobi/TDF/FTC RAL+TDF/FTC
  NNRTI-Based Regimens:
  EFV plus ABC/3TC or RPV/TDF/FTC
  PI-Based Regimen:
  ATV/r plus ABC/3TC
  PI-Based Regimens:
  DRV/r + ABC/3TC or LPV/r + ABC/3TC or LPV/r + TDF/FTC
  INSTI-Based Regimen:
  RAL plus ABC/3TC
  And other ART regimens
  EFV/TDF/FTC: standard combination therapy
  ATV/r + TDF/FTC or DRV/r + TDF/FTC
  DTG+ABC/3TC DTG+TDF/FTC EVG/cobi/TDF/FTC RAL+TDF/FTC
  EFV plus ABC/3TC or RPV/TDF/FTC
  ATV/r plus ABC/3TC
  DRV/r + ABC/3TC or LPV/r + ABC/3TC or LPV/r + TDF/FTC
  RAL plus ABC/3TC
  Other ART regimens
Period: Overall Study
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B) | Group 2 Standard Combination Therapy
Started | 49 | 25
Completed | 47 | 20
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Population: Baseline measures are reported for the 74 participants who initiated treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B) | Group 2 Standard Combination Therapy | Total
Number analyzed (Participants) | 49 | 25 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 50 (13) | 50 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 4 | 16
  Male | 37 | 21 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 49 | 24 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Free of Therapeutic Failure
Description: Proportion of patients free of therapeutic failure at week 24. Therapeutic failure includes virological failure, change in treatment for any reason, consent withdrawal, loss to follow-up or death
Time Frame: 24 weeks
Population: A total of 75 subjects were randomized. However, in the RAL/3TC group (n=50), one subject was excluded due to consent withdrawal prior to the initiation of medication and therefore did not complete the Baseline (randomization) visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 49 | 25
Participants
  No events | 47 | 20
  Lost to follow up | 0 | 2
  Pregnancy | 1 | 0
  Stops treatment | 0 | 2
  Virological faiulure | 0 | 1
  Stops study medical decision | 1 | 0

2. Secondary Outcome: Efficacy in Virological Suppression Assessed With Ultrasensitive HIV-1 RNA Detection (Limit of Detection 1 Copy/mL)
Time Frame: 24 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Changes in Peripheral Mononuclear Blood Cells HIV-1 Reservoir
Time Frame: 24 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Insulin Resistance (HOMA-IR)
Description: Composite measure
Time Frame: 24 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Changes in Body Fat Composition
Description: Composite measure
Time Frame: 24 weeks
Population: Some patients were not performed a DEXA during the study
Measure: Mean (Standard Deviation); unit: percentage of fat weight
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 46 | 25
percentage of fat weight
  Baseline extremities fat percentage | 54.13 (19.44) | 49.43 (21.26)
  Baseline total fat percentage | 28.50 (7.62) | 27.54 (8.75)
  Week 24 extremities fat percentage: number analyzed (Participants) | 44 | 20
  Week 24 extremities fat percentage | 54.09 (17.68) | 50.21 (23.77)
  Week 24 total fat percentage: number analyzed (Participants) | 44 | 20
  Week 24 total fat percentage | 28.84 (7.23) | 28.78 (9.55)

6. Secondary Outcome: Changes in Plasma 25-OH Vitamin D Levels
Time Frame: 24 weeks
Population: Some patients vitamine D determination was not available
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 45 | 24
ng/mL
  Baseline | 17.4 (9.0) | 16.7 (9.6)
  week 24: number analyzed (Participants) | 45 | 19
  week 24 | 29.5 (15.1) | 26.5 (17.2)

7. Secondary Outcome: Changes in Estimated Glomerular Filtration Rate (CKD-EPI)
Description: Composite measure
Time Frame: 24 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Changes in CD38
Time Frame: 24 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Changes in IL-6
Time Frame: 24 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Changes in Sleep Quality (Pittsburgh Sleep Quality Index)
Description: The Pittsburgh Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven áreas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month.
  The posible range of the scale is from 0 to 21 points. The greater the score the poorest is the sleep quality.
Time Frame: 24 weeks
Population: Some patients did not complete the questionnaire
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 46 | 22
score on a scale
  Baseline score | 5 (3.5) | 4.7 (3.1)
  Week 24 score: number analyzed (Participants) | 38 | 18
  Week 24 score | 4.8 (3.1) | 5.1 (3.5)

11. Secondary Outcome: Changes in Adherence in Both Treatment Arms (Morisky-Green Test)
Description: Patients were asked to complete the Morisky-Green questionnaire:
  Some people forget to take their medication as prescribed. How often does it happen to you? (Always/often/sometimes/rarely/never) Some people forget some taking of the medication or change the prescribed schedule / take to adapt it to their own needs. How often do you do it? (Always/often/sometimes/rarely/never) Some people stop taking their medications as prescribed when they feel better. How often do you do it? (Always/often/sometimes/rarely/never) Some people stop taking their medications as prescribed when they feel worse. How often do you do it? (Always/often/sometimes/rarely/never)
  Only if patients answered never to each four questions, they were considered adherent; if not, non adherent.
Time Frame: 24 weeks
Population: Some patients did not complete the questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 49 | 25
Participants
  Baseline: Adherent | 19 | 11
  Baseline: Non adherent | 29 | 13
  Baseline: Not evaluated/ Lost follow Up | 1 | 1
  Week 24: Adherent | 19 | 14
  Week 24: Non adherent | 27 | 5
  Week 24: Not evaluated/ Lost follow Up | 3 | 6

12. Secondary Outcome: Changes in Total Cholesterol
Time Frame: 24 weeks
Population: Some patients have not performed all the protocol determinations
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 49 | 25
mg/dl
  Baseline | 189 (46) | 187 (44)
  Week 24: number analyzed (Participants) | 47 | 19
  Week 24 | 190 (45) | 186 (37)

13. Secondary Outcome: Changes in HDL Cholesterol
Time Frame: 24 weeks
Population: Some patients did not performed all the determinations
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 49 | 25
mg/dl
  Baseline | 48 (15) | 46 (13)
  Week 24: number analyzed (Participants) | 47 | 19
  Week 24 | 49 (14) | 45 (15)

14. Secondary Outcome: Changes in LDL Cholesterol
Time Frame: 24 weeks
Population: Some patients did not perform all the determinations
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 45 | 22
mg/dl
  Baseline: number analyzed (Participants) | 44 | 22
  Baseline | 120 (39) | 115 (29)
  Week 24: number analyzed (Participants) | 45 | 19
  Week 24 | 119 (40) | 118 (33)

15. Secondary Outcome: Changes in Triglycerides
Time Frame: 24 weeks
Population: All patients did not perform all the determinations
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 49 | 25
mg/dl
  Baseline | 98.5 (49.9) | 112.0 (53.0)
  Week 24: number analyzed (Participants) | 47 | 19
  Week 24 | 97.7 (44.8) | 100.9 (37.3)

16. Secondary Outcome: Changes in Bone Mineral Density
Description: DEXA
Time Frame: 24 weeks
Population: Not all the patients performed the DEXA
Measure: Mean (Standard Deviation); unit: gr/cm^2
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 47 | 25
gr/cm^2
  Baseline | 1166.1 (100.9) | 1211.6 (79.6)
  Week 24: number analyzed (Participants) | 43 | 19
  Week 24 | 1183.0 (98.5) | 1247.4 (80.9)

17. Secondary Outcome: Changes in Urine Beta-2-microglobulin/Creatinine Ratio
Time Frame: 24 weeks
Population: Some patients did not performed this determination
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B | Group 2 Standard Combination Therapy
Number analyzed (Participants) | 19 | 7
mg/g
  Baseline | 672.8 (773.3) | 595.3 (948.7)
  Week 24: number analyzed (Participants) | 9 | 4
  Week 24 | 275.7 (227.2) | 788.5 (1587.3)

18. Secondary Outcome: Changes in HLA-DR
Time Frame: 24 weeks
Reporting Status: Not Posted

19. Secondary Outcome: Changes in High Sensitivity C-reactive Protein
Time Frame: 24 weeks
Reporting Status: Not Posted

20. Secondary Outcome: Changes in Mononuclear Activation SD-14
Time Frame: 24 weeks
Reporting Status: Not Posted

21. Secondary Outcome: Changes in Mononuclear Activation SD-163
Time Frame: 24 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: An adverse event (AE) is any untoward occurrence to the health of a patient or clinical trial subject treated with a medicinal product and which does not necessarily have a causal relationship with this treatment.
  A total of 75 subjects were randomized. However, in the RAL/3TC group (n=50), one subject was excluded due to consent withdrawal prior to the initiation of medication and therefore did not complete the Baseline (randomization) visit.
Groups:
- Group 1 Raltegravir / 3TC (MK0518B): Raltegravir / 3TC (MK0518B ) (50 patients)
  Raltegravir/3TC: MK0518B (Raltegravir/3TC) (300mg/150mg) twice daily, administered orally in the 300/150 mg film-coated tablets according to instructions in the prescribing information.
Arm/Group | Group 1 Raltegravir / 3TC (MK0518B) | Group 2 Standard Combination Therapy
All-Cause Mortality (participants affected / at risk) | 1/49 | 0/25
Serious Adverse Events (participants affected / at risk) | 3/49 | 3/25
Other Adverse Events (participants affected / at risk) | 12/49 | 10/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Raltegravir / 3TC (MK0518B) (N=49) | Group 2 Standard Combination Therapy (N=25)
Altered blood test (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — On May 30, 2016 goes to the emergency room. In the analysis we can see elevation of ldh, ck, anemia and thrombocytopenia not present in previous analyzes so it is admitted for study.
Prostate Neoplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Patient with well-controlled hiv infection. Suspected prostate neoplasia (biopsy due to thrombocytopenia) with bone metastasis, metastatic medullary infiltration
hilar adenopathies and anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — hilar adenopathies and anemia
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — disseminated melanoma
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — umbilical hernia, inguinal hernia
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
febrile syndrome (Infections and infestations) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — 3-day course of diarrhea
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Raltegravir / 3TC (MK0518B) (N=49) | Group 2 Standard Combination Therapy (N=25)
Amigdalitis (Infections and infestations) | 3 (3) | 1 (1)
Ansiety (Psychiatric disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Insomnia (Psychiatric disorders) | 4 (4) | 0 (0)
Lues (Infections and infestations) | 1 (1) | 3 (3)
Dizziness (Gastrointestinal disorders) | 3 (3) | 1 (1) — Sickness or emesis
Common cold (Infections and infestations) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-11-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT02284035/Prot_SAP_000.pdf